CLINICAL TRIAL: NCT01937130
Title: A Placebo-Controlled, Multicenter, Double-Blind, Randomized, Pharmacokinetic and Pharmacodynamic Trial of IDN-6556 in Subjects With Acute-on-Chronic Liver Failure
Brief Title: Pharmacokinetic and Pharmacodynamic Study of IDN-6556 in ACLF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data needs met
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDN-6556-02
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Acute on Chronic Hepatic Failure; Acute Liver Failure; Liver Cirrhosis; Acute Alcoholic Hepatitis
Keywords: Liver Failure; Cirrhosis; Alcoholic Hepatitis
MeSH Terms: conditions — Liver Failure, Acute; Liver Cirrhosis; Liver Failure; Fibrosis; Hepatitis, Alcoholic | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IDN-6556 5 mg (Experimental): Dosed twice daily
  Interventions: Drug: IDN-6556
- IDN-6556 25 mg (Experimental): Dosed twice daily
  Interventions: Drug: IDN-6556
- IDN-6556 50 mg (Experimental): Dosed twice daily
  Interventions: Drug: IDN-6556
- Placebo (Placebo Comparator): Dosed twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IDN-6556
  Other Names: emricasan; PF-03491390
  Arms: IDN-6556 25 mg; IDN-6556 5 mg; IDN-6556 50 mg
Other: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the pharmacokinetics, pharmacodynamics, safety and preliminary efficacy of IDN-6556 in subjects with cirrhosis of the liver who are hospitalized for more than 24 hours due to acute deterioration of liver function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and understand and comply with the requirements of the study
* Subjects with a clinical, radiological and/or histological diagnosis of cirrhosis
* Subjects having not required hospital admission within 4 weeks of screening for a complication of cirrhosis
* Subjects with an acute deterioration of liver function
* Subjects who meet one of the following criteria:

  1. Subjects with renal failure (defined as creatinine ≥ 2.0 to ≤ 3.4 mg/dL)
  2. Subjects with other single organ failure with i. Renal impairment (defined as an increase in creatinine of > 0.3 mg/dL from either an established prior Baseline level or if applicable, upon admission to hospital if prior level is unavailable; for inclusion, the creatinine level must be raised above normal levels), and/or ii. Hepatic encephalopathy grade I or II
  3. Subjects with two organ failures
* If a subject received steroids for alcohol-induced acute liver failure, he/she must be unresponsive to steroid therapy. Responsiveness is based on investigator discretion.
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from screening to one month after the last dose of study drug

Exclusion Criteria:

* Known infection with HIV
* Subjects with cirrhosis who develop decompensation at any time in the postoperative period following partial hepatectomy
* Subjects with evidence of uncontrolled infection defined as persistent bacterial culture positivity despite adequate antibiotic therapy
* Subjects with clinical evidence of disseminated intravascular coagulation
* Subjects with chronic and/or pre-existing kidney disease defined as eGFR (estimated glomerular filtration rate) of less than 30 mL/min for 3 months or longer
* Subjects who are hypotensive (defined as mean arterial pressure <70 mmHg) or require the use of inotropic support
* Subjects with evidence of significant and/or uncontrolled bleeding
* Subjects requiring mechanical ventilation
* Subjects with active or history of malignancies other than hepatocellular carcinoma (HCC) within Milan criteria or curatively treated skin cancer (basal cell or squamous cell carcinomas), unless adequately treated or in complete remission for five or more years
* Subjects previously exposed to IDN-6556
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QT or QTc interval of > 480 milliseconds (msec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ryder, Dr., Principal Investigator — Nottingham University Hospital NHS Trust
Locations (26):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Scripps Clinic, La Jolla, California
  - VA San Diego Healthcare System, San Diego, California
  - Sutter Pacific Medical Foundation, San Francisco, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Univerisity of Louisville Liver Research Center, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Montefiore Medical Center, The Bronx, New York
  - University of Utah, Salt Lake City, Utah
  - University of Washington Harborview Medical Center, Seattle, Washington
- United Kingdom (15):
  - Singleton Hospital, Swansea, Wales
  - Basildon and Thurrock University Hospital, Basildon
  - Blackpool Victoria Hospital, Blackpool
  - Bristol Royal Infirmary, Bristol
  - Ninewells Hospital, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - University College London, Royal Free Hospital, London
  - Royal London Hospital, London
  - Central Manchester University Hospitals NHS Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 33 subjects were screened at 14 sites, and 23 subjects were randomized to one of the 4 treatment arms.
Pre-assignment Details: 23 subjects were randomized but 21 subjects received treatment. 1 subject lost due to death and 1 subject lost due to withdrew of consent. 7 subject of 21 completed the treatment phase (Day 28). 4 of 3 completed the two follow-up phone calls made at Months 3 and 6. 14 subjects discontinued the study early.
Groups:
- IDN-6556 5 mg; IDN-6556 25 mg; IDN-6556 50 mg: Dosed twice daily
  IDN-6556
- Placebo: Dosed twice daily
  Placebo
Period: Overall Study
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo
Started | 5 | 7 | 5 | 4
Completed | 0 | 3 | 2 | 2
Not Completed | 5 | 4 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1
Not completed — Death | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Patients unable to swallow | 0 | 1 | 0 | 0
Not completed — Patient lost to FU due to death | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with acute-on-Chronic liver failure (ACLF)
Groups:
- Total: Total of all reporting groups
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo | Total
Number analyzed (Participants) | 5 | 7 | 5 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 4 | 4 | 20
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49.0 [41 to 60] | 50.0 [30 to 58] | 61.0 [42 to 71] | 53.5 [34 to 59] | 50.0 [30 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 3 | 5 | 3 | 2 | 13
Region of Enrollment [Number; unit: participants]
  United States | 0 | 2 | 1 | 2 | 5
  United Kingdom | 5 | 5 | 4 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC)
Description: Primary endpoints for AUC_0-8, AUC_0 last, AUC_0-inf on Day 1 and Day 4 for the active treatment arms were analyzed.
Time Frame: 28 days
Population: AUC_0-last: The number of participants analyzed in the 25mg arm was 7 at Day 1 AUC_0-inf: The number of participants analyzed in the 5mg arm was 2 at Day 1 and 0 at Day 4, in the 25mg arm was 5 at Day 1 and 2 at Day 4, in the 50mg arm was 2 at Day 1 and 3 at Day 4.
  Values listed as "0" were non-estimable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Units Other Than Participants: Number of Participants Analyzed at Day 4
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg
Number analyzed (Participants) | 5 | 5 | 5
Number analyzed (Number of Participants Analyzed at Day 4) | 4 | 4 | 5
h*ng/mL
  Day 1 AUC 0-8 | 275 (40.0) | 1165 (45.3) | 2397 (99.3)
  Day 4 AUC 0-8 | 224.3 (36.9) | 1767 (31.4) | 2148 (227.9)
  Day 1 AUC 0-last | 275 (40.0) | 1295 (33.4) | 2997 (103.8)
  Day 4 AUC 0-last | 224.3 (36.9) | 1818 (27.8) | 2294 (257.9)
  Day 1 AUC 0-inf | 0 (0) | 1462 (30.3) | 0 (0)
  Day 4 AUC 0-inf | 0 (0) | 0 (0) | 3447 (188.2)

2. Primary Outcome: Cmax
Description: Primary endpoints forCmax on Day 1 and Day 4 for the active treatment arms were analyzed.
Time Frame: 28 Days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng/mL)
Units Other Than Participants: Number of Participants Analyzed at Day 4
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg
Number analyzed (Participants) | 5 | 7 | 5
Number analyzed (Number of Participants Analyzed at Day 4) | 4 | 5 | 5
(ng/mL)
  Day 1 Cmax | 84.4 (43.9) | 329.8 (48.3) | 696.1 (117.4)
  Day 4 Cmax | 38.0 (33.9) | 586.5 (33.7) | 594.1 (161.3)

3. Primary Outcome: Tmax & t1/2 Parameters
Description: Primary endpoints for tmax & t1/2 on Day 1 and Day 4 for the active treatment arms were analyzed.
Time Frame: 28 Days
Population: t1/2 number of participants analyzed at Day 1 in the 5mg arm was 2 and 1 at Day 4, in the 25mg arm was 5 at Day 1 and 2 at Day 4, in the 50mg arm was 2 at Day 1 and 3 at Day 4.
  Values listed as "0" were non-estimable values.
Measure: Mean (Standard Deviation); unit: (h)
Units Other Than Participants: Number of Participant Analyzed at Day 4
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg
Number analyzed (Participants) | 5 | 7 | 5
Number analyzed (Number of Participant Analyzed at Day 4) | 4 | 5 | 5
(h)
  Day 1 tmax | 3.0 (1.3) | 2.9 (1.5) | 3.6 (3.0)
  Day 4 tmax | 3.8 (3.4) | 2.7 (1.8) | 3.5 (2.8)
  Day 1 t1/2 | 0 (0) | 2.2 (0.7) | 0 (0)
  Day 4 t1/2 | 0 (0) | 0 (0) | 3.4 (2.7)

4. Secondary Outcome: Levels of CK18/M30
Description: Caspase-cleaved cytokeratin serum levels (CK18/M30)
Time Frame: Baseline, Day 2, Day 4, Day 7, Day 14, Day 21, and Day 28
Population: Number of subjects analyzed varied by time point; Day2: 5 and 25 arms are 4 and 6; Day4: 25 and placebo arms are 6 and 2; Day7: 25 arm is 6; Day14: 5, 25, 50, and placebo arms are 2, 5, 3, and 2; Day21: 5, 25, 50, and placebo arms are 2, 3, 2, and 2; Day28: 5, 25, 50, and placebo arms are 0, 3, 2, and 2; "0" are non-estimable values
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo
Number analyzed (Participants) | 5 | 7 | 5 | 3
U/L
  Baseline | 703 [302 to 2162] | 1392 [330 to 3593] | 919 [395 to 1851] | 455 [240 to 1716]
  Day 2 | 465 [323 to 1999] | 616 [277 to 2162] | 348 [179 to 1023] | 425 [284 to 1496]
  Day 4 | 717 [427 to 2162] | 847 [306 to 2016] | 362 [237 to 822] | 634 [297 to 970]
  Day 7 | 562 [331 to 2162] | 1226 [326 to 1993] | 319 [203 to 2985] | 466 [278 to 1388]
  Day 14 | 1307 [452 to 2162] | 1149 [325 to 2071] | 577 [521 to 954] | 843 [317 to 1369]
  Day 21 | 850 [222 to 1478] | 770 [298 to 1512] | 551 [341 to 760] | 626 [297 to 955]
  Day 28 | 0 [0 to 0] | 808 [386 to 975] | 533 [186 to 879] | 553 [214 to 892]

5. Secondary Outcome: Levels of CK18/M65
Description: Caspase full-length cytokeratin serum levels CK18/M65
Time Frame: Baseline, Day 2, Day 4, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo
Number analyzed (Participants) | 5 | 7 | 5 | 3
U/L
  Baseline | 1345 [876 to 2862] | 2819 [277 to 3762] | 1946 [705 to 6999] | 1324 [507 to 2451]
  Day 2 | 1058 [702 to 3145] | 2116 [157 to 3155] | 1287 [665 to 4365] | 1195 [531 to 2213]
  Day 4 | 1237 [1100 to 2664] | 2257 [783 to 3033] | 1436 [662 to 4566] | 990 [548 to 1431]
  Day 7 | 1364 [751 to 3098] | 2601 [733 to 6999] | 1997 [695 to 4028] | 1086 [614 to 1948]
  Day 14 | 1961 [893 to 3028] | 3067 [1027 to 5971] | 1286 [1010 to 3711] | 1310 [686 to 1934]
  Day 21 | 3809 [619 to 6999] | 2039 [400 to 3502] | 2500 [987 to 4012] | 1125 [721 to 1529]
  Day 28 | 0 [0 to 0] | 1825 [654 to 1845] | 2119 [532 to 3705] | 1027 [500 to 1553]

6. Secondary Outcome: Levels of Caspase 3/7 RLU
Description: Concentration of Caspase 3/7 Relative Light Units
Time Frame: Baseline, Day 2, Day 4, Day 7, Day 14, Day 21, and Day 28
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: RLU
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo
Number analyzed (Participants) | 5 | 7 | 5 | 3
RLU
  Baseline | 4418 [2516 to 6692] | 3967 [2615 to 6884] | 4304 [1135 to 5405] | 4074 [3189 to 5331]
  Day 2 | 2893 [2222 to 6268] | 1487 [842 to 3071] | 974 [653 to 1323] | 3989 [3934 to 4078]
  Day 4 | 3147 [1479 to 6025] | 1136 [741 to 15674] | 1204 [657 to 4253] | 5853 [5778 to 5928]
  Day 7 | 4081 [979 to 5611] | 1271 [636 to 3794] | 958 [603 to 1390] | 3917 [2672 to 5269]
  Day 14 | 2265 [1214 to 3315] | 1180 [434 to 1623] | 835 [276 to 897] | 1869 [1273 to 2465]
  Day 21 | 2914 [1948 to 3880] | 636 [471 to 1105] | 962 [833 to 1091] | 1590 [970 to 2210]
  Day 28 | 0 [0 to 0] | 1208 [679 to 2949] | 963 [859 to 1066] | 1894 [874 to 2914]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for a period of 18 months.
Arm/Group | IDN-6556 5 mg | IDN-6556 25 mg | IDN-6556 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 3/5 | 6/7 | 3/5 | 2/4
Other Adverse Events (participants affected / at risk) | 3/5 | 7/7 | 4/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDN-6556 5 mg (N=5) | IDN-6556 25 mg (N=7) | IDN-6556 50 mg (N=5) | Placebo (N=4)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDN-6556 5 mg (N=5) | IDN-6556 25 mg (N=7) | IDN-6556 50 mg (N=5) | Placebo (N=4)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Cardiac disorders (Cardiac disorders) | 1 | 1 | 0 | 0
Eye disorders (Eye disorders) | 0 | 1 | 1 | 0
Gastrointestinal disorders (Gastrointestinal disorders) | 3 | 7 | 4 | 3
General disorders and administration site conditions (General disorders) | 1 | 3 | 2 | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 2 | 3 | 1 | 1
Infections and infestations (Infections and infestations) | 1 | 2 | 1 | 0
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Investigations (Investigations) | 1 | 1 | 0 | 3
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Nervous system disorders (Nervous system disorders) | 2 | 4 | 2 | 0
Psychiatric disorders (Psychiatric disorders) | 1 | 2 | 1 | 0
Renal and urinary disorders (Renal and urinary disorders) | 0 | 0 | 2 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 2
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Vascular disorders (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less